CLINICAL TRIAL: NCT04846257
Title: Specific Preoperative Dynamic Contrast-enhanced MRI Semi-quantitative Markers Can Correlate With Vascularity in Specific Areas of the Glioblastoma Tissue and Predict Recurrence
Status: Completed | Type: Observational
Sponsor: Egyptian Medical Syndicate (Other)
Responsible Party: Principal Investigator, Mohammed A. Azab, Principal Investigator, Cairo University
Other Study IDs: DCE_MRI_GBM
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dynamic contrast-enhanced MRI — Dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) is the acquisition of sequential images during the passage of a contrast agent within a tissue of interest.

SUMMARY:
Radiological Markers of vascularity as wash-in rate, washout rate, and capillary time to peak in different single tumour regions were extracted for all glioblastoma patients before being surgically resected from preoperative DCE-MRI. Tissue samples were obtained from different intratumoral regions and peritumoral oedema and evaluated for the vascular endothelial growth factor (VEGF)

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed glioblastoma with a maximum diameter from 3-5 cm as a single lesion identified by MRI.
* The lesions should be surgically resected at the time of the presentation.

Exclusion Criteria: N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed glioblastoma
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Recurrence of tumor | 2018-2021

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Cairo University Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided